CLINICAL TRIAL: NCT04926545
Title: Mechanistic and Pharmacokinetic Studies of Classical Chinese Formula Xiao Chai Hu Tang Against Irinotecan-Induced Gut Toxicities(Clinical Study Part:Run-in Safety Study)
Brief Title: XCHT for Irinotecan-Induced Gut Toxicities (Run-in Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: University of Houston (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021KT1005; 81961128028 (Other Grant/Funding Number: National Nature Science Fundation of China)
Record Dates: First submitted 2021-05-30; First posted 2021-06-15 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-04

CONDITIONS: Malignant Tumor; Diarrhea
Keywords: Malignant tumor; Irinotecan; chemotherapy-induced diarrhea; Classical Chinese Formula; safety
MeSH Terms: conditions — Neoplasms; Diarrhea | interventions — shosaiko-to; Long-Term Synaptic Depression; Raloxifene Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irinotecan naive cohort (Experimental): This cohort will enroll 6 postmenopausal female patients who have never received irinotecan treatment before. Patients in irinotecan naive cohort will receive 3 cycles of FOLFIRI chemotherapy, during which 4 rounds of pharmacokinetic studies will be conducted.
  Round 0 (before chemotherapy): pharmacokinetic testing (raloxifene 60mg as probe) before XCHT administration, then XCHT for 4 days with pharmacokinetic testing (raloxifene 60mg as probe) on the 4th day of XCHT administration.
  Round 1(1st cycle of chemotherapy): XCHT for 5 days and FOLFIRI on day 4, with pharmacokinetic testing (without raloxifene) on day 4.
  Round 2 (2nd cycle of chemotherapy): XCHT for 5 days and FOLFIRI on day 4, with pharmacokinetic testing (raloxifene 60mg as probe) on day 3.
  Round 3 (3rd cycle of chemotherapy): XCHT for 5 days and FOLFIRI on day 4, with pharmacokinetic testing (raloxifene 60mg as probe) on day 3.
  Interventions: Drug: Xiao Chai Hu Tang (XCHT); Other: Raloxifene; Drug: FOLFIRI regimen
- Irinotecan used cohort (Experimental): This cohort will recruit 18 patients who were treated with irinotecan previously and have at least one diarrhea episode with a severity of more than grade 2. Patients in irinotecan used cohort will receive 3 cycles of FOLFIRI chemotherapy, during which 3 rounds of pharmacokinetic studies will be conducted.
  Round 1(1st cycle of chemotherapy): FOLFIRI, with pharmacokinetic testing (raloxifene 60mg as probe) on the first day of chemotherapy.
  Round 2 (2nd cycle of chemotherapy): XCHT for 5 days and FOLFIRI on day 4, with pharmacokinetic testing (raloxifene 60mg as probe) on day 4.
  Round 3 (3rd cycle of chemotherapy): XCHT for 5 days and FOLFIRI on day 4, with pharmacokinetic testing (raloxifene 60mg as probe) on day 3.
  Interventions: Drug: Xiao Chai Hu Tang (XCHT); Other: Raloxifene; Drug: FOLFIRI regimen

INTERVENTIONS:
Drug: Xiao Chai Hu Tang (XCHT) — XCHT 9g, po qd, 3 days before each cycle of chemotherapy for 5 days, except the 1st cycle of chemotherapy for irinotecan used cohort patients.
  Additional XCHT, 9g qd will be orally administrated for 4 days during the Round 0 study for irinotecan naive cohort patients.
  Other Names: Xiao Chai Hu Tang granules from Nin Jiom Medicine Manufactory (Hong Kong) Ltd.
Other: Raloxifene — Raloxifene 60mg po, used as probe for pharmacokinetic testing. For irinotecan naive cohort patients, raloxifene 60mg will be orally administrated on Day 1 and Day 5 (4th day of XCHT administration) during round 0 study, Day 3 (the day before chemotherapy) during round 2 and round 3 study. For irinotecan used cohort patients, raloxifene 60mg will be orally administrated on Day 1 (irinotecan using day) during round 1 study, Day 4 (irinotecan using day) during round 2 study, and Day 3 (the day before chemotherapy) during round 3 study.
  Other Names: Evista from Eli Lilly
Drug: FOLFIRI regimen — Patients will receive 3 cycles of FOLFIRI regimen for chemotherapy. Irinotecan intravenous (IV) infusion (180 mg/m2) through a drip into the bloodstream over 90 minutes. Folinic acid (400 mg/m2) IV infusion through a drip into the bloodstream over 2 hours. 5-fluorouracil (5-FU) IV bolus (400 mg/m2) into the bloodstream over 5 minutes, followed by 5-FU (2400 mg/m2) continuous IV infusion through a drip or pump into the bloodstream for 46-48 hours.
  Other Names: Irinotecan Hydrochloride from Pfizer+Folinic acid+5-fluorouracil (5-FU)

SUMMARY:
Run-in safety study, to determine the safety of co-administration of irinotecan, raloxifene, and Xiao Chai Hu Tang (XCHT), and to optimize the blood collection time points for pharmacokinetic (PK) study for another randomized control trial.

DETAILED DESCRIPTION:
There will be two cohorts with a total of 24 patients in this study. Cohort A will enroll 6 naïve postmenopausal female patients who have never received irinotecan treatment before. Patients in this group will have 4 rounds of studies following different protocol to determine (1) the impact of XCHT on raloxifene PK (Round 0, co-administration of XCHT and raloxifene); (2) the impact of XCHT on irinotecan PK (Round 1, co-administration of XCHT and standard FOLFIRI); (3) the safety of co- administration of XCHT, raloxifene, and FOLFIRI and evaluation of raloxifene as a probe for XCHT treatment to prevent irinotecan-induced severe delayed-onset diarrhea (Round 2 and 3, co-administration of XCHT, raloxifene, and standard FOLFIRI). The reason to recruit postmenopausal women is that these patients usually take raloxifene to prevent osteoporosis and the risk of raloxifene is expected to be limited.

Cohort B will recruit 18 patients who were treated with irinotecan previously and have at least one diarrhea episode with a severity of ≥grade 2. The reason we propose to recruit patients who had diarrhea induced by irinotecan is that these patients are supposed to be sensitive to irinotecan so that we can determine the PK changes and safety. Patients in this group will have 3 rounds of FOLFIRI chemotherapy to determine (1) the impact of FOLFIRI on raloxifene PK (Round 1, co-administration of FOLFIRI with raloxifene); (2) the complete PK profile of SN-38, SN-38G, raloxifene, raloxifene-glucuronide, and XCHT components (Round 2, co- administration of FOLFIRI with XCHT and raloxifene); and (3) the safety of co-administration of XCHT, raloxifene, and FOLFIRI in sensitive patients and evaluation of raloxifene as a probe for XCHT treatment to prevent irinotecan-induced diarrhea (Round 3, co-administration of XCHT, raloxifene and standard FOLFIRI).

ELIGIBILITY:
Cohort A: Naïve (no irinotecan treatment before) postmenopausal female cancer patients.

Inclusion criteria:

1. Malignant tumor confirmed by histology or cytology;
2. Postmenopausal women, after bilateral oophorectomy; age > 60 years old, or age < 60 years old with menopause for more than 1 year;
3. Age ≥ 18 years old, ≤ 75 years old;
4. ECOG score of the patient ≤ 2 points;
5. Never been treated with irinotecan;
6. Plan to receive at least 3 rounds of FOLFIRI chemotherapy determined by physicians;
7. Normal organ functions can meet the requirements for systemic chemotherapy:

   * Reserve functions of normal bone marrow: absolute neutrophil count (ANC) ≥ 1.5×109/L, PLT ≥ 100×109/L, hemoglobin ≥ 90 g/L;
   * Normal renal functions: serum creatinine ≤ 1.5 mg/dl (133 μmol/L) and/or creatinine clearance ≥ 60 ml/min;
   * Normal hepatic functions: total serum bilirubin level ≤ 1.5 times of the upper limit of normal value (ULN), serum aspartate aminotransferase (AST) & alanine aminotransferase (ALT) ≤ 2.5 × ULN; If abnormal hepatic functions are caused by a potentially malignant tumor, and AST ＆ ALT ≤ 5 × ULN;
8. Patient is willing to participate and cooperate to complete the questions in the case report form;
9. Patient can understand and sign the informed consent form, is well compliant, and can be followed up.

Cohort B: cancer patients who experienced irinotecan -induced diarrhea (grade >2)

Inclusion criteria:

1. Malignant tumor confirmed by histology or cytology;
2. Age ≥ 18 years old, ≤ 75 years old;
3. ECOG score of the patient ≤ 2 points;
4. Patients who have diarrhea worse than grade 2 due to irinotecan chemotherapy (the last dose of irinotecan is administered within 1 month);
5. Patients who plan to receive 3 rounds of FOLFIRI chemotherapy;
6. Normal organ functions can meet the requirements for systemic chemotherapy:

   * Reserve functions of normal bone marrow: absolute neutrophil count (ANC) ≥ 1.5×109/L, PLT ≥ 100×109/L, hemoglobin ≥ 90g/L;
   * Normal renal functions: serum creatinine ≤ 1.5mg/dl (133μmol/L) and/or creatinine clearance ≥ 60ml/min;
   * Normal hepatic functions: total serum bilirubin level ≤ 1.5 times of the upper limit of normal value (ULN), serum aspartate aminotransferase (AST) & alanine aminotransferase (ALT) ≤ 2.5 × ULN; If abnormal hepatic functions are caused by a potentially malignant tumor, and AST ＆ ALT ≤ 5 × ULN;
7. Patient is willing to participate and cooperate to complete the questions in the case report form;
8. Patients can understand and sign the informed consent form, is well compliant, and can be followed up.

Exclusion Criteria:

1. Patients with diagnosed depression, obsession or/and schizophrenia;
2. Patients with diagnosed inflammatory bowel diseases (including Crohn's disease, ulcerative colitis)
3. Patient with active tuberculosis and other uncontrolled infections;
4. Patient has previously received radiotherapy on the abdominal cavity and pelvic cavity;
5. Pregnant or lactating women;
6. Patient previously had or is now having thromboembolic (blood clotting) events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Average trajectory of irinotecan, raloxifene, XCHT and their metabolites (14 compounds) | The blood samples (2.0 ml) will be collected at 8 points for each Round (hour 0, hour 0.5, hour 1, hour 2, hour 4, hour 6, hour 8, and hour 24 after raloxifene administration)
  Plasma concentration for each compounds will be tested at 8 points for each Round.

SECONDARY OUTCOMES:
incidences of grade ≥3 diarrhea | Through study completion, an average of 2 months
  The diarrhea severity will be evaluated following standard criteria in NCI-CTC AE 5.0
occult blood test for stool | Through study completion, an average of 2 months
  occult blood test for stool, reported as negative, weak positive, and positive.
incidence of other chemo-related adverse effects | Through study completion, an average of 2 months.
  Other adverse reactions will be evaluated following standard criteria in NCI-CTC AE 5.0
incidence of diarrhea (grade ≥2) | Through study completion, an average of 2 months.
  The diarrhea severity will be evaluated following standard criteria in NCI-CTC AE 5.0 Grade 2 is defined as Stool is increased by 4-6 times each day relative to baseline; discharge from stoma moderately increased.

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Zhang, Prof, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No